CLINICAL TRIAL: NCT01842594
Title: A Phase II Trial of Combined Hydroxychloroquine and Sirolimus in Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Most patients completed only the primary objective (PET) and not went throught the secondary outcome (efficacy phase) of 8wks period.
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120306M
Record Dates: First submitted 2012-12-19; First posted 2013-04-29 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Sarcoma
Keywords: Sarcoma, Hydroxychloroquine, Sirolimus, PET
MeSH Terms: conditions — Sarcoma | interventions — Sirolimus; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus and hydroxychloroquine (Experimental): Both hydroxychloroquine 200 mg/tab and sirolimus 1 mg/tab are pills each are taken 2 tablet orally once daily(QD) for 2 cycles . Each treatment cycle is 28 days.
  Interventions: Drug: Sirolimus and hydroxychloroquine

INTERVENTIONS:
Drug: Sirolimus and hydroxychloroquine — Both hydroxychloroquine 200 mg/tab and sirolimus 1 mg/tab are pills each are taken 2 tablet orally QD for 2 cycles .
  Each treatment cycle is 28 days.

SUMMARY:
Determine the objective response rate in sarcoma patients treated with hydroxychloroquine and sirolimus.

DETAILED DESCRIPTION:
This study evaluates the daily morning single dose of hydroxychloroquine /sirolimus combined therapy in sarcoma patients. Study arm were treated with hydroxychloroquine 400 mg /sirolimus 2mg gd for 8-wk therapy. Patients will be discontinued from the study after 8-wk observation period.

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study.

TREATMENT PLAN:

1. Both hydroxychloroquine 200 mg/tab and sirolimus 1 mg/tab are pills each are taken 2 tablet orally every day. Treatment will be divided into time periods called cycles. Each treatment cycle is 28 days. The exception to this 28 day cycle is when participants start taking the pills for the first time. When the hydroxychloroquine and sirolimus begins, the first cycle of 28 days begins.
2. There are several tests and procedures that will be performed at specific time periods during protocol treatment. These include: blood work, performance status assessment, questions about medical history and medications, tumor assessment with PET/CT or MRI and, eye exams.
3. Dose modification criteria:

Participants may continue to receive study treatment as long as they experienced grade 1 or 2 side effects. The treatment drug will be 50% reduction of dose in any grade 3 toxicity; and discontinued of treatment (off-study) in any grade 4 toxicity or disease progression during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Soft tissue sarcoma (including high grade or low grade soft tissue sarcoma、osteogenic sarcoma and the following 4 recurrent benign tumors which may have aggressive clinical course after initial surgical treatment : lymphangioleiomyomatosis、angiomyolipoma、giant cell tumor、phylloid tumor) that are refractory to at least first line full course of standard chemotherapy, relapsed after standard chemotherapy, or who have no standard therapy available and refused chemotherapy
* Patients must be >/= 21 years.
* Patients must be >/= 4 weeks beyond treatment with a cytotoxic chemotherapy regimen, or therapeutic radiation, or major surgery. Patients may have received palliative localized radiation immediately before or during treatment provided that radiation is not delivered to the only site of disease being treated under this protocol. For biologic/targeted agents patients must be >/= 5 half-lives or >/= 3 weeks form the last dose (whichever comes first).
* Eastern Cooperative Oncology Group(ECOG) performance status </= 2
* Patients must have certain organ and marrow function resave defined as: White blood cell(WBC_ >/= 3,000/mL;platelets >/=100,000/mL; creatinine </= 2 X Upper Limit of Normal (ULN); total bilirubin </= 2.0; Alanine Aminotransferase(ALT;SGPT) </= 5 X ULN; Exception for patients with liver metastasis: total bilirubin </= 3 x ULN; ALT(SGPT) </= 8 X ULN;cholesterol </= 350 mg/dL; triglycerides </= 400 mg/dL (sirolimus and hydroxychloroquine only).
* Patients must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

* Uncontrolled intercurrent illness, including, but not limited to, uncontrolled infection, uncontrolled asthma, need for hemodialysis, need for ventilatory support.
* Pregnant or lactating women.
* History of hypersensitivity to sirolimus.
* History of hypersensitivity to hydroxychloroquine
* Patients unwilling or unable to sign informed consent document.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Chi MS, Lee CY, Huang SC, Yang KL, Ko HL, Chen YK, Chung CH, Liao KW, Chi KH. Double autophagy modulators reduce 2-deoxyglucose uptake in sarcoma patients. Oncotarget. 2015 Oct 6;6(30):29808-17. doi: 10.18632/oncotarget.5060. PMID 26375670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between August 2012 and June 2014 at Department of Radiation Therapy and Oncology, Shin Kong Wu Ho-Su Memorial Hospital.
Groups:
- Sirolimus and Hydroxychloroquine: Patients received 1 mg of sirolimus (rapamycin, Rapa) and 200 mg of hydroxychloroquine (HCQ) twice a day before a meal for 2 weeks.
Period: Overall Study
Arm/Group | Sirolimus and Hydroxychloroquine
Started | 13
Completed | 10
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Sirolimus and Hydroxychloroquine: Patients received 1 mg of Rapa and 200 mg of HCQ twice a day before a meal for 2 weeks.
Arm/Group | Sirolimus and Hydroxychloroquine
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 63 [17 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Standardized Uptake Values (SUVmax) Change on PET/CT Scan
Description: A baseline whole-body [18F]-fluorodeoxyglucose(FDG) PET was performed before therapy initiation. Patients received 1 mg of Rapa and 200 mg of HCQ twice a day before a meal for 2 weeks. A second [18F]-FDG PET was performed after treatment completion. SUVs were calculated for all lesions. Regions of interest (ROI) were contoured to represent tumors (>2 cm) and organs (lungs, spleen, and liver) on all transaxial and coronal slices. ROIs were normalized for injection dose and body weight, and the maximum voxel value was recorded for each region or organ. The highest SUV measured with increased uptake was considered the SUVmax. Correlative diagnostic CT examinations were used for accurate localization of the lesions. The most intense uptake at baseline was identified as the index lesion and evaluated for treatment response.
Time Frame: 2 Weeks
Measure: Mean (95% Confidence Interval); unit: percentage of the SUVmax Change
Units Other Than Participants: lesions
Arm/Group | Sirolimus and Hydroxychloroquine
Number analyzed (Participants) | 10
Number analyzed (lesions) | 34
percentage of the SUVmax Change | -19.6 [-30.1 to -9.1]

2. Secondary Outcome: The Toxicity
Description: Number of Participants with Adverse Events. Toxicities parameters are according to the Nation Cancer Institute Common Terminology Criteria for Adverse Event, version 3.0.
Time Frame: 2 Weeks
Measure: Number; unit: participants
Arm/Group | Sirolimus and Hydroxychloroquine
Number analyzed (Participants) | 10
participants | 3

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Sirolimus and Hydroxychloroquine
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus and Hydroxychloroquine (N=10)
Skin rash (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes